CLINICAL TRIAL: NCT02975453
Title: Study of Risk Factors of Major Cardiovascular Events in Patients With Nonvalvular Atrial Fibrillation Treated With a Direct Oral Anticoagulant (Rivaroxaban)
Brief Title: Study of Major Cardiovascular Events in Patients With Nonvalvular Atrial Fibrillation Treated With Rivaroxaban
Acronym: EMIR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18884
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban: Non-valvular atrial fibrillation (NVAF) patients treated with rivaroxaban for at least 6 months prior to the study inclusion
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by the treating physician

SUMMARY:
Evaluation of the performance of the 2MACE index in a population of nonvalvular atrial fibrillation (NVAF) patients treated with rivaroxaban in Spain

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients with diagnosis of NVAF.
* Patients treated with rivaroxaban from at least six months prior to the study inclusion.
* Patients who have been given appropriate information about the study objectives and procedures and who have given their written informed consent.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Patients who initiate treatment with rivaroxaban after the start of the study inclusion period.
* Prosthetic heart valves or the presence of any severe valvulopathies.
* Patients with severe cognitive impairment.
* Patients with chronic infections (HIV infection, hepatitis C virus, hepatitis B virus) or systemic autoimmune diseases.
* Patients with active cancer.
* Patients with liver insufficiency (eg. cirrhosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-valvular atrial fibrillation who are under rivaroxaban treatment and that attend the Cardiology Units at Spanish hospitals and private clinics
Sampling Method: Non-Probability Sample
Enrollment: 1481 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
2MACE score | At baseline
  MACE: Major adverse cardiovascular events. 2MACE: History of Myocardial infarction/ Cardiac revascularization and Metabolic Syndrome, Age >75 years, Congestive heart failure (ejection fraction <40%), Thrombo-Embolism
Occurrence of MACE to evaluate the performance of the 2MACE index | At 2 years and 6 months or early termination
  Percentage of patients with MACE including fatal/nonfatal myocardial infarction, cardiac revascularization and cardiovascular death

SECONDARY OUTCOMES:
Incorporation of additional risk factors to the 2MACE index or replacing some of the existing ones | At baseline
  Risk factors to the 2MACE index (e.g. body mass index, smoking, drugs use, estimated glomerular filtration rate, structural cardio-pathology)
Occurrence of major cardiovascular events (fatal/nonfatal myocardial infarction, cardiac revascularization and cardiovascular death) | At baseline, at 1 year, at 2 years, at 2 years and 6 months or early termination
Occurrence of stroke | At baseline, at 1 year, at 2 years, at 2 years and 6 months or early termination
Occurrence of transient ischemic attack (TIA) | At baseline, at 1 year, at 2 years, at 2 years and 6 months or early termination
Occurrence of systemic embolism | At baseline, at 1 year, at 2 years, at 2 years and 6 months or early termination
Thromboembolic risk based on the CHADS2 score | At baseline
  CHADS2: Cardiac Failure, Hypertension, Age, Diabetes, Stroke
Thromboembolic risk based on the CHA2DS2-VASC | At baseline
  CHA2DS2-VASc:Cardiac failure, Hypertension, Age ≥75, Diabetes, Stroke -Vascular disease, Age and Sex category
Number of MACEs occurring during the study | At 1 year, at 2 years, at 2 years and 6 months or early termination
Patients' profile | At baseline
  Baseline patients' profile defined by: sociodemographic data, anthropometric data, previous relevant medical history, cardiac medical history distinct to atrial fibrillation, comorbidities (renal failure, left ventricular dysfunction, hypertension, thyroid dysfunction, liver failure, alcoholism)
Number of cases (frequency) of metabolism syndrome at enrollment with/without the occurrence of myocardial infarction or coronary revascularization | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Spain

REFERENCES:
- [Background] Rivera-Caravaca JM, Anguita Sanchez M, Sanmartin Fernandez M, Rafols C, Baron-Esquivias G, Arribas Ynsaurriaga F, Freixa-Pamias R, Lekuona Goya I, Vazquez Rodriguez JM, Perez-Cabeza AI, Cosin-Sales J, Urena Montilla I, Alvarez-Vieitez Blanco A, Marin F. Adverse Clinical Outcomes and Associated Predictors in Rivaroxaban-Treated Atrial Fibrillation Patients With Renal Impairment. Am J Cardiol. 2023 Sep 15;203:122-127. doi: 10.1016/j.amjcard.2023.06.105. Epub 2023 Jul 22. PMID 37487406
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/